CLINICAL TRIAL: NCT05243927
Title: Comparison of Aerobic Exercise and Spinal Stabilization Exercises in Women With Primary Dysmenorrhea
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ankara Yildirim Beyazıt University (Other)
Responsible Party: Principal Investigator, seyda toprak celenay, associate professor, Ankara Yildirim Beyazıt University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022/02/08
Record Dates: First submitted 2022-02-08; First posted 2022-02-17 (Actual); Last update posted 2022-02-17 (Actual); Status verified 2022-02

CONDITIONS: Primary Dysmenorrhea

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic exercise group (Experimental): Aerobic exercise will be performed under the supervision of a physiotherapist with a treadmill during 40-60 minutes, 3 days a week for 8 weeks.
  Interventions: Other: Aerobic exercise program
- Stabilization exercise group (Active Comparator): Spinal stabilization exercises will be performed with a physiotherapist during 40-60 minutes, 3 days a week for 8 weeks.
  Interventions: Other: Spinal stabilization exercise program

INTERVENTIONS:
Other: Aerobic exercise program — Aerobic exercise will be performed under the supervision of a physiotherapist with a treadmill during 40-60 minutes 3 days a week for 8 weeks
  Arms: Aerobic exercise group
Other: Spinal stabilization exercise program — Spinal stabilization exercises will be performed with a physiotherapist during 40-60 minutes 3 days a week for 8 weeks.
  Arms: Stabilization exercise group

SUMMARY:
The aim of the study is to compare the effects of aerobic exercise and spinal stabilization exercises in women with primary dysmenorrhea (PD) complaints.

DETAILED DESCRIPTION:
PD is the cramping pain that comes before or during a period. Different exercise approaches have positive effects in PD. Comparing the effects of these exercise approaches is needed to determine the effects on PD.

ELIGIBILITY:
Inclusion Criteria:

Women with primary dysmenorrhea complaint according to the Primary Dysmenorrhea Consensus Guide, Over 18 years of age, Having a mean pain intensity of moderate and higher according to the Visual Analogue Scale in the last 6 months, Having a regular menstrual cycle (28±7 days), Volunteered to participate in the study.

Exclusion Criteria:

Having a pathological history and radiological findings pointing to secondary dysmenorrhea, Using oral contraceptives/antidepressants at least 6 months, Receiving hormone therapy, Undergoing pelvic surgery, Pregnant, Giving birth, Using an intrauterine device, Having neurological, orthopedic and/or rheumatological diseases Having a history of ischemic heart disease (recently myocardial infarction, angina pectoralis, uncontrolled hypertension, etc.), Having a psychiatric disease, Having a history of malignancy

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Primary dysmenorrhea is a gynecological problem that can be seen in most women.
Enrollment: 40 (Estimated)
Dates: Start 2022-03 (Estimated); Primary Completion 2023-03 (Estimated); Study Completion 2023-08 (Estimated)

PRIMARY OUTCOMES:
Menstrual pain intensity | change from baseline at 8 weeks
  Menstrual pain intensity will be evaluated with Visual Analogue Scale. This scale consists of a 10 cm horizontal line. The starting point "0" = "no pain", while "10" = "unbearable pain". Individuals will be asked to mark on a 10 cm straight line according to the level of pain they feel. Pain intensity will be recorded by measuring the distance between the beginning of the line and the marked place.

SECONDARY OUTCOMES:
Menstrual symptoms | change from baseline at 8 weeks
  Menstrual symptoms will be measured with the menstrual symptom questionnaire. Menstrual Symptom Questionnaire is a 24-item self-report scale and each item is scored between 1 (never) and 5 (always). An increase in the mean score indicates an increase in the severity of menstrual symptoms. The total score is 120 points.
Impacts of academic/work performance | change from baseline at 8 weeks
  Impacts of academic/work performance will be evaluated with Visual Analogue Scale. This scale consists of a 10 cm horizontal line. The starting point "0"= means "my work/school performance is not affected in any way", while "10"= means "my work/school performance is greatly affected".
Impacts of life quality | change from baseline at 8 weeks
  Impacts of life quality will be evaluated with Visual Analogue Scale. This scale consists of a 10 cm horizontal line. The starting point "0" = "my quality of life is not affected in any way", while "10" = "my quality of life is greatly affected". Individuals will be asked to mark on a 10 cm straight line according to the quality of life they think.
Functional and emotional effects | change from baseline at 8 weeks
  Functional and emotional effects will be evaluated with Functional and Emotional Dysmenorrhea Scale. Options in the 14-item scale are (1) not at all similar to my situation, (2) Not similar to my situation, (3) Both similar and not similar to my situation, (4) considered similar to my situation, (5) very similar to my situation. The total score range is between 14-70. As the scores obtained from the scale increase, the functional and emotional state of being affected by dysmenorrhea also increases.
Sleep quality | change from baseline at 8 weeks
  Sleep quality will be evaluated with Jenkins Sleep Scale, which consists of 4 items. Each item is rated with a 6-point Likert Scale. The total score ranges from 0 to 20. An average of at least 4 or more is considered a sleep quality disorder.
Trunk muscle endurances | change from baseline at 8 weeks
  Trunk muscle endurances will be evaluated with McGill's endurance tests. During the tests, individuals will be asked to maintain the determined positions and the elapsed time will be recorded in seconds. The test result is recorded in seconds.
Posture | change from baseline at 8 weeks
  Posture will be evaluated with PostureScreen Mobile application. PostureScreen Mobile application is an application that evaluates posture anterior-posterior-lateral photographically and provides data by comparing deviations that can be seen in posture according to ideal standing posture.
Pelvic tilt | change from baseline at 8 weeks
  Pelvic tilt will be evaluated with Palpation Meter (PALM) device. The PALM device is an inclinometer and a palpation meter consisting of two caliper arms, which are used to measure the lumbopelvic position and pelvic tilt.
Functional capacity | change from baseline at 8 weeks
  Functional capacity will be evaluated with a 2 kilometer walking test. The time taken for walking is calculated by substituting the heart rate, body mass index and age at the end of walking. The result obtained is evaluated according to age and gender, and an appropriateness index is found.
Subjective perception of improvement | After exercise program (at 8 week)
  Subjective perception of improvement will be evaluated with 4-item Likert-type scale (worse, same, better, improved).

CONTACTS AND LOCATIONS:
Overall Officials: Seyda Toprak Celenay, Principal Investigator — Ankara Yildirim Beyazıt University